CLINICAL TRIAL: NCT07367763
Title: The Relationship Between Self-Awareness and Risk of Falls During Walking in Adults From Rehabilitation Settings and the Community
Brief Title: The Relationship Between Self-Awareness and Risk of Falls During Walking in Adults
Acronym: SAFR
Status: Active, not recruiting | Type: Observational
Sponsor: University of Haifa (Other)
Collaborators: Clalit Health Services (Other)
Responsible Party: Principal Investigator, Galit Yogev-Seligmann, Senior Lecturer, Department of Physical Therapy, Faculty of Social Welfare and Health Sciences, University of Haifa, University of Haifa
Other Study IDs: COM2-0046-22_076-25; COM2-0046-22 (Other: Helsinki Committee, Clalit Health Services)
Record Dates: First submitted 2025-09-25; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Falls; Fall Risk; Fall Risk Factors; Cognitive Dysfunction; Self-Awareness; Gait Disorders
Keywords: Self-Awareness; Falls; Fall Risk; Dual-Task Walking; Executive Function; Gait; Older Adults; Rehabilitation; Cognitive Function
MeSH Terms: conditions — Cognitive Dysfunction; Mobility Limitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults: Adults aged 60-85 living in the community, ambulatory independently or with a cane

SUMMARY:
This study examines the relationship between self-awareness and the risk of falls during walking in older adults and rehabilitation patients. Falls are a major health concern among older adults worldwide. Many studies have shown that executive functions, such as attention and problem-solving, are related to fall risk; however, little is known about the role of self-awareness-the ability to recognize one's own strengths, limitations, and errors-in predicting falls.

In this study, approximately 100 participants (adults aged 60-85 years) will be recruited from both a rehabilitation day center and community settings. Participants will complete cognitive tests, self-awareness questionnaires, and walking assessments using wearable sensors. Walking will be tested both at a normal pace and while performing a secondary task (dual-task walking).

The results will help clarify whether reduced self-awareness is an independent risk factor for falls. Findings may improve fall-prevention strategies in both rehabilitation and community settings.

The study protocol has been reviewed and approved by the Faculty Ethics Committee, University of Haifa, and the Helsinki Committee of Clalit Health Services.

DETAILED DESCRIPTION:
Falls are among the most common health issues in older adults, with 30-40% of individuals aged 65 and older experiencing at least one fall each year. Falls are strongly associated with reduced quality of life, increased healthcare costs, and higher mortality rates. Executive dysfunction has consistently been identified as a major predictor of fall risk. Yet impaired self-awareness-defined as the ability to accurately evaluate one's own abilities, limitations, and errors-has rarely been studied as an independent risk factor.

The present study is designed to examine whether reduced self-awareness contributes uniquely to fall risk in adults. It combines two cohorts under one protocol: (1) patients recruited from a day rehabilitation center, and (2) community-dwelling older adults. All particpants will undergo identical assessments.

Study outcome measures

* Montreal Cognitive Assessment (MoCA) for global cognition (also a screening test for cognitive decline)
* NeuroTrax™ computerized executive function and attention tests
* Phonemic Verbal Fluency (PVF) task
* Patient Competency Rating Scale (PCRS) and task-specific awareness questionnaires
* Gait analysis using APDM Mobility Lab™ sensors under single-task (normal walking) and dual-task (walking + PVF) conditions

This observational, cross-sectional study will recruit approximately 100 participants (from rehabilitation and from the community). Inclusion criteria: age 60-85 years, Hebrew or Arabic speakers, ambulatory independently or with a cane, and living with a spouse or caregiver who can provide informant data. Exclusion criteria: medical diagnoses significantly affecting cognition or ambulation, hospitalization within the last month, and MoCA score below 20.

The findings are expected to expand the understanding of fall risk factors by highlighting the role of self-awareness. Results may inform future interventions and clinical guidelines for fall prevention in both clinical and community populations.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60-85 years
* Men and women
* Ambulatory independently or with a cane
* Hebrew or Arabic speakers, able to read and write
* Living with a spouse or caregiver who can provide informant questionnaire data

Exclusion Criteria:

* Medical diagnosis significantly affecting cognition, emotion, or ambulation
* Hospitalization within the past month
* Montreal Cognitive Assessment (MoCA) score below 20

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community-dwelling older adults and patients attending a rehabilitation day center, all aged 60-85 years, who are ambulatory independently or with a cane and able to complete cognitive and awareness assessments.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Competency Rating Scale (PCRS-2) Discrepancy Score | baseline
  Self-awareness will be assessed using the Patient Competency Rating Scale (PCRS-2), which includes both self-report and proxy-report forms. The outcome measure will be the discrepancy score between patient and caregiver ratings, reflecting the participant's level of awareness across cognitive, emotional, social, and functional domains.
Gait Speed and Variability | baseline
  Gait performance will be objectively measured using APDM Mobility Lab sensors. Primary gait parameters include walking speed (m/s) and step-to-step variability (%). Dual-task cost will be calculated as the relative change in gait parameters between single-task and dual-task walking, serving as indicators of gait stability and fall risk.

SECONDARY OUTCOMES:
Self-Awareness Walking Questionnaire Score | baseline
  Participants will complete a short questionnaire rating their perceived walking stability and safety under single-task (normal walking) and dual-task (walking while performing a cognitive task) conditions. The outcome measure will be the mean score across items, reflecting task-specific self-awareness.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Haifa, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet certain whether individual participant data (IPD) will be shared. The decision will depend on future publication requirements, institutional guidelines, and participant privacy considerations.